CLINICAL TRIAL: NCT00313430
Title: Urinary Concentration and Diluting Ability in Patients With Chronic Renal Disease or Hypertension
Brief Title: Urinary Concentration and Diluting Ability in Patients With Chronic Renal Disease and/ or Hypertension
Status: Completed | Type: Observational
Sponsor: Erling Bjerregaard Pedersen (Other)
Responsible Party: Sponsor-Investigator, Erling Bjerregaard Pedersen, professor, chief physician, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Other Study IDs: MED. RES.HOS 2004 03/IT
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Renal Insufficiency, Chronic; Hypertension
Keywords: Urine concentration ability; chronic renal insufficiency; hypertension; aquaporin2; Patients with chronic renal insufficiency; Patients with hypertension; Healthy volunteers
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Dialysis patients
- with or wthout glucose added to dialysis fluid

SUMMARY:
The investigators want to test the hypothesis that patients with chronic renal disease have a poorer ability to preserve water after being thirsty and a poorer ability to excrete water after a load of fluid. They presume that these abilities become poorer when renal insufficiency progresses. The investigators further hypothesize that patients with hypertension also have a decreased ability to concentrate and dilute urine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal insufficiency, aged between 18 and 65, both men and women
* Creatinine clearance between 30-59 ml/min
* Patients with hypertension, aged between 18 and 65, both men and women; hypertension is defined as a mean arterial blood pressure in the daytime that is more than 140/90 mm Hg.
* Healthy volunteers, aged between 18 and 65, both men and women

Exclusion Criteria:

* Clinical signs or history of disease in the heart, lungs, liver, brain, and endocrine organs
* Cancer
* Alcohol abuse
* Medicine abuse
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy participants were recruited by advertisements in public and private institutions Patients with primary hypertension or chronic renal failure were recruited from the Out-patients' Clinic, Department of Medicine, Section of Nephrology, Holstebro Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2004-05; Primary Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Holstebro, Holstebro, Denmark
Locations (1):
- Department of Medicine, Holstebro Hospital, Holstebro, Ringkjoebing, Denmark

REFERENCES:
- [Derived] Pedersen EB, Thomsen IM, Lauridsen TG. Abnormal function of the vasopressin-cyclic-AMP-aquaporin2 axis during urine concentrating and diluting in patients with reduced renal function. A case control study. BMC Nephrol. 2010 Oct 5;11:26. doi: 10.1186/1471-2369-11-26. PMID 20923561